CLINICAL TRIAL: NCT01189942
Title: A Phase 1b Study of FOLFIRI Plus OMP-21M18 as 1st or 2nd-line Treatment in Subjects With Metastatic Colorectal Cancer
Brief Title: A Study of FOLFIRI Plus OMP-21M18 as 1st or 2nd-line Treatment in Subjects With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M18-003
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Cancer
Keywords: Phase 1; dose escalation; histologically; confirmed; malignancy; metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — demcizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: OMP-21M18 — The first 6 participants will receive OMP21M18 2.5 mg/kg once every other week, the next 6 participants will receive 5 mg/kg once every other week, and the final 6 participants will receive 10 mg/kg once every other week. A Data Safety Monitoring Board (DSMB) will review the data for the 6 participants in each dose level after the last participant in that group has been treated for 56 days and decide whether it is safe to move up to the next highest dose level. After confirming the optimum dose, 14 additional participants will be treated at the highest dose level that the DSMB considers safe.

SUMMARY:
The purpose of this study is to test the safety and determine the optimal dose of a new drug, OMP-21M18, when given in combination with FOLFIRI, a standard drug treatment for advanced colorectal cancer. Participants must not have had more than one chemotherapy regimen for their metastatic disease. OMP-21M18 is a humanized monoclonal antibody (a protein made in the laboratory) developed to target cancer stem cells. The way the body handles OMP-21M18 will also be investigated.

Up to 32 participants, 21 years or older, at up to 6 centres in Australia and New Zealand, will receive intravenous infusions of OMP-21M18 followed by FOLFIRI every two weeks, until disease progression or limited by drug toxicity. After 8 weeks, participants will undergo assessments to determine their disease status. If there is no evidence of disease progression participants will continue to receive infusions of OMP-21M18 and FOLFIRI every second week, until disease progression.

DETAILED DESCRIPTION:
Current cancer therapies often produce an initial reduction in tumour size but may not have longterm benefits. One possible explanation for this is the presence cancer cells known as a cancer stem cells. Cancer stem cells represent a small part of the tumour but are believed to be responsible for much of the growth and spread of the cancer. They may also be more resistant to traditional types of therapy, such as chemotherapy and radiation therapy.

The purpose of this study is to test the safety and determine the optimal dose of a new experimental drug, OMP-21M18, when given in combination with FOLFIRI, a chemotherapy regimen consisting of the following three medications: folinic acid (leucovorin), 5fluorouracil and irinotecan. The administration of these three medications is a standard treatment for advanced colorectal cancer. OMP-21M18 is a humanized monoclonal antibody (a protein made in the laboratory) developed to target cancer stem cells. The way the body handles OMP21M18 will also be investigated.

Up to 32 participants, 21 years or older, will be enrolled at up to 6 centres in Australia and New Zealand. Following informed consent and screening, FOLFIRI will be administered once every 14 days (or until toxicity necessitates reducing or delaying a dose). OMP-21M18 will be administered by intravenous (IV) infusion once every 14 days on the same day as FOLFIRI. A Data Safety Monitoring Board (DSMB) will review the data for the 6 participants in each dose level after the last participant in that group has been treated for 56 days and decide whether it is safe to move up to the next highest dose level. After confirming the optimum dose, 14 additional participants will be treated at the highest dose level that the DSMB considers safe.

Participants will be assessed for disease status every 8 weeks and for safety at every visit and for 30 days after the end of study drug treatment. Safety will be assessed by adverse event monitoring, physical examination, vital signs, blood tests, cardiac monitoring, and participant interview. Response rates, duration of response, time to progression, and survival will be evaluated requiring CT or MRI scans and CEA (tumour marker) levels at baseline and then every 8 weeks. The development of antibodies to treatment will be assessed throughout the study and up to 12 weeks after the end of study drug treatment. During the study blood samples will be taken to assess whether OMP21M18 is producing desired changes to the genes and proteins related to the cancer (biomarkers). The study includes an optional part which will investigate how variations in people's genetic makeup affect their response to medications. This involves the collection of one blood sample just before participants receive their first dose of study treatment. DNA will be extracted from the blood sample for testing.

ELIGIBILITY:
Inclusion criteria

1. Subjects must have histologically confirmed metastatic colorectal cancer. Subjects may not have received more than 1 prior chemotherapy regimen for their metastatic disease and may not have received irinotecan for treatment of their metastatic disease.
2. Age >21 years
3. ECOG performance status <2 (see Appendix B)
4. Life expectancy of more than 3 months
5. Subjects must have normal organ and marrow function as defined below:

   * Leukocytes >3.5 x 109/L
   * Absolute neutrophil count >1.25 x 109/L
   * Hemoglobin >100 g/L
   * Platelets >125 X 109/L
   * Total bilirubin <2 X institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) <5 X institutional ULN
   * Alkaline phosphatase <5 X institutional ULN
   * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) within institutional ULN
   * Creatinine <1.5 X institutional ULN OR
   * Calculated creatinine clearance >60 mL/min using the Cockcroft and Gault formula as follows:

   Creatinine clearance (mL/min) = (140 - age) x ideal body weight [kg] 0.814 x serum creatinine [µmol/L] For women multiply the value from the equation above by 0.85. Where age is in years, weight is in kg, and serum creatinine is in µmol/L
6. Women of childbearing potential must have had a prior hysterectomy or have a negative serum pregnancy test and be using adequate contraception prior to study entry and must agree to use adequate contraception from study entry through at least 6 months after discontinuation of study drug. Men must also agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and from study entry through at least 6 months after discontinuation of study drug. Should a woman enrolled in the study or a female partner of a man enrolled in the study become pregnant or suspect she is pregnant while participating in this study or within 6 months after discontinuation of study drug, the Investigator should be informed immediately.
7. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria

Subjects who meet any of the following criteria will not be eligible for participation in the study:

1. Subjects receiving any other investigational agents or anti-cancer therapy.
2. Subjects with brain metastases (subjects must have a CT scan or MRI of the head within 28 days prior to enrollment to rule out brain metastases), uncontrolled seizure disorder, or active neurologic disease
3. History of a significant allergic reaction attributed to humanized or human monoclonal antibody therapy
4. Significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
5. Pregnant women or nursing women
6. Subjects with known HIV infection
7. Known bleeding disorder or coagulopathy
8. Subjects receiving heparin, warfarin, or other similar anticoagulants. Note: Subjects may be receiving low-dose aspirin and/or non-steroidal anti-inflammatory agents.
9. Subjects with known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease
10. New York Heart Association Classification II, III, or IV (See Appendix D)
11. Subjects with a blood pressure of >140/90 mmHg. The BP should be taken using the method described in Section 9.3. Subjects taking antihypertensive medications must be taking ≤ 2 medications to obtain this level of BP control.
12. Subjects with tumors that are currently involving the lumen of the gastrointestinal tract
13. Subjects with current evidence of cardiac ischemia or heart failure within the last 6 months, subjects who are receiving any medications for cardiac ischemia, subjects with a B-type natriuretic peptide (BNP) value of >200 pg/mL, subjects with a LVEF < 45%, or subjects that have received a total cumulative dose of ≥400 mg/m2 doxorubicin.
14. Subjects with ECG evidence of ischemia or ≥ Grade 2 ventricular arrhythmia, subjects who have a history of acute myocardial infarction within 6 months, or subjects with unstable angina.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To the determine the maximum tolerated dose of OMP-21M18 plus FOLFIRI | Will be done after each patient in dose cohort reaches Day 56

SECONDARY OUTCOMES:
To determine the safety of FOLFIRI plus OMP-21M18 at two dose levels | Until disease progression plus 30 days after
To determine the rates of immunogenicity of FOLFIRI plus OMP-21M18 | Up until 12 weeks after patient has Disease Progression
To determine population pharmacokinetics | Until Disease Progression
To determine the exploratory biomarker changes of FOLFIRI plus OMP 21M18 | Until Disease Progression
To determine the preliminary efficacy of FOLFIRI plus OMP-21M18 | Until Disease Progression

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (4):
  - Sydney Cancer Centre, Camperdown, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Waikato Hospital, Hamilton, New Zealand